CLINICAL TRIAL: NCT06565338
Title: Comparison Between the Neuroprotective Effect of Vitamin D Versus Dexmedetomidine in Patients with Traumatic Brain Injury Using Interleukin 6 As Inflammatory Marker
Brief Title: Comparison Between Effect of Vitamin D Versus Dexmedetomidine in Patients with Head Trauma Using Interleukin 6
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, asmaa elhelw, Investigator, Minia University
Other Study IDs: 403
Record Dates: First submitted 2024-07-30; First posted 2024-08-21 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Dexmedetomidine; Cholecalciferol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- group A: dexmedetomidine 0.4 mic/kg loading dose then 0.25 mic/kg/hr for 5 days
  Interventions: Drug: Dexmedetomidine
- group B: vitamin D 100.000 IU given IM once
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Dexmedetomidine — drug
  Other Names: precedex
  Groups: group A
Drug: Vitamin D3 — drug
  Other Names: depovit - decaprino
  Groups: group B

SUMMARY:
in this study the investigators compare between the neuroprotective effect of vitamin d versus dexmedetomidine in patients with traumatic brain injury using interleukin 6 as inflammatory biomarker

DETAILED DESCRIPTION:
patients with moderate head trauma (GCS 8-12) within first 24 hours were randomly divided into 2 groups, first group received 100,000 IU of vitamin D was given IM & the other group received dexmedetomidine 0.4 mic/kg as loading dose then 0.25 mic/kg/hr as maintainence dose for 5 days detecting APATCHE at admission and following up of vital signs (HR & NIBP) & investigations (CBC & RFT& ABG & ESR& CRP & IL-6) & GCS and GOS for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Both Gender.
* Age (18-50)
* GCS (8-12)
* Pt with traumatic brain insult who not indicated surgical intervention

Exclusion Criteria:

* Prior severe disability.
* Isolated brain system lesions.
* History of underlying neurologic, metabolic or psychiatric disorders.
* Alcohol or drug abuse.
* Pregnancy.
* Patients with intracranial hemorrhage who indicated surgical evacuation.
* Multisystem life-threatening trauma.
* GCS > 12 & <8.
* Vitamin d deficiency.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with traumatic brain injury with GCS 8-12
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint aims to measure the inflammatory markers level: | 5 days
  1- IL-6 in the unit of (pg/mL).
Primary outcome measure | 5 days
  2- ESR in the unit of(mm/hr).
Primary outcome measure | 5 days
  3- CRP in the unit of (mg/L).

SECONDARY OUTCOMES:
The secondary endpoints aim to compare ICU stay, morbidity and mortality in both groups: | 3 months
  1- ICU stay (no. Of days)
Secondary outcome measure | 3 month
  2- Glascow outcome scale (1-5) : that determine morbidity and mortality (units on scale from 1 to 5 with better scale towards 5 and worse towards 1)

CONTACTS AND LOCATIONS:
Overall Officials: ahmed ezz, Study Chair — Minia University
Locations (1):
- Asmaa, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No